CLINICAL TRIAL: NCT03131752
Title: Early Pulmonary Rehabilitation With Elastic Resistance in Exacerbated COPD Patients
Brief Title: Early Pulmonary Rehabilitation in Exacerbated COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Valeria Amorim Pires Di Lorenzo, PhD, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ElastRes COPD 2016
Record Dates: First submitted 2017-03-30; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; muscle strength; physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The patients will be evaluated on 4 phases: at the first contact (at least 24 hours after drug therapy and at most 48 hours), 7 days, 30 days and 3 months after the first contact. They will be submitted to an anamnesis, assessment of muscular strength, physical activity level, functional capacity, dyspnea on activity daily living and quality of life.
  The intervention will last 7 days for all the patients. Three phases will be performed: warm up, knee muscle strengthening with elastic bands and stretch/relax.
  Interventions: Behavioral: Elastic Resistance Intervention in Exacerbated Patients
- Control Group (No Intervention): The patients will be evaluated on 4 phases: at the first contact (at least 24 hours after drug therapy and at most 48 hours), 7 days, 30 days and 3 months after the first contact. They will be submitted to an anamnesis, assessment of muscular strength, physical activity level, functional capacity, dyspnea on activity daily living and quality of life.
  Patients will be not receive intervention.

INTERVENTIONS:
Behavioral: Elastic Resistance Intervention in Exacerbated Patients — The intervention protocol will performed during 7 days for all patients and this will begin 24 -48 hours after the start of medication for exacerbation. Those who are hospitalized and discharged before this period will continue their treatment at the Laboratory of Spirometry and Respiratory Physiotherapy (LEFIR) of the Federal University of São Carlos. The intervention will also perform for at least 5 continuous days. The ideal elastic band for the training will be chosen through the test of 10 maximum repetitions. The test and the training will be performed in an ergonomic chair allowing the lower limbs to remain pending. After 24 hours of the test, patients will perform knee extension exercise with the appropriate elastic band. Three sets of 10 repetitions will be done in each exercise, with a minimum rest interval of 1 minute between sets or until heart rate values return to baseline. Patients will be re-evaluated 1 and 3 months after the first contact.
  Other Names: GI
  Arms: Intervention Group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by chronic and progressive airflow limitations and subjects with COPD also experience exacerbations characterized by the worsening of respiratory symptoms. It's necessary medical intervention, changes in regular medication, and the use of antibiotics and/or corticosteroids followed or not by hospitalization. The exacerbations contribute to worsening of the disease with systemic impairment and muscle weakness is a very relevant event. The physical inactivity, especially related to bed rest, comprises one of the factors contributing to muscle atrophy and loss of muscle strength. Thus, the intervention performed during hospitalization is necessary to minimize the consequences which causes impairment in health status subjects. The aim of the study is assess the effect of the intervention with elastic bands, in muscle strength,level of the physical activity, functional capacity, dyspnea on activities of daily living (ADL) and quality of life in COPD exacerbation subjects. Moreover,verify the intervention benefits over 01 and 03 months post exacerbation episode. It will be a prospective, randomized, longitudinal and interventional study. The investigators will be asses both gender patients with exacerbation of COPD in 4 situations: First time (at least 24 and at most 48 hours after the beginning of medical therapy); seven days post the first assessment; one and three months post exacerbation episode. It will be assess the muscle strength, physical activity level, functional capacity, dyspnea on ADL and quality of life. The patients will be randomized in 2 groups: intervention and control group. The intervention will be performed with elastic bands once a day during seven days. The investigators expected that patients of the intervention group will present better muscle strength, physical activity level and functional capacity than the control group. Furthermore, an improvement in dyspnea and quality of life is expected in intervention group when compared as with control group patients. It is hypothesized that the benefits of intervention will be maintained over one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or more, of both genders, who are in a an exacerbation of the disease according to Global Initiative for Chronic Obstructive Lung Disease (GOLD,2015) refered by the doctors, hospitalized or not in exacerbation treatment .All patients should be in spontaneous breathing at the time of assessment, in oxygen use or not and in conditions to understand the proposed evaluations; Patients who use non-invasive ventilation will also be included as long as it does not interfere with the protocols; All should agree to participate in the research in a free and informed manner. Patients who are referred to the Intensive Care Unit (ICU) may be included 24 hours after discharge from the ICU.

Exclusion Criteria:

* Patients who present with orthopedic limitations, other pulmonary diseases, rheumatological, cardiovascular or neurological disorders that not allow the assessment. Patients whit drug os alcohol dependence, patients undergoing invasive mechanical ventilation, hemodynamic instability, the presence of unstable angina, will be excluded. In addition, patients with cognitive deficits that impair comprehension of the assessments will be excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-06-07 (Estimated); Primary Completion 2017-08-07 (Estimated); Study Completion 2019-03-07 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength pre and post first contact | 24-48 hours after the start of exacerbation medication and 7 days after the first contact
  The effect of intervention or no intervention on muscle strength will be evaluated by the portable dynamometer (Microfet 2®, Hoggan - Health Industries, West Jordan, UT, USA). It will be positioned in front of the leg to assess quadriceps strength.
Muscle Strength Follow-up | 1 month after the first contact
  The benefits of intervention or no intervention on muscle strength will be evaluated by the portable dynamometer (Microfet 2®, Hoggan - Health Industries, West Jordan, UT, USA).It will be positioned in front of the leg to assess quadriceps strength 1 month after the first contact.
Muscle Strength Follow-up 2 | 3 months after the first contact
  The muscle strength 3 months after exacerbation will be evaluated by the portable dynamometer (Microfet 2®, Hoggan - Health Industries, West Jordan, UT, USA). It will be positioned in front of the leg to assess quadriceps strength 3 months after the first contact.

SECONDARY OUTCOMES:
Physical activity level pre and post first contact | 24-48 hours after the start of exacerbation medication and 7 days after the first contact
  The effect of intervention or no intervention on physical activity level will be evaluated by the actigraph (activPAL3TM - PAL Technologies Ltd., Glasgow, United Kingdom) through the number of steps, time spent in different positions during 7 days.
Physical activity level Follow-up | 1 month after the first contact
  The benefits of intervention or no intervention on physical activity level will be evaluated by the actigraph (activPAL3TM - PAL Technologies Ltd., Glasgow, United Kingdom) through the number of steps, time spent in different positions during 7 days, 1 month after the first contact.
Physical activity level Follow-up 2 | 3 months after the first contact
  The physical activity level 3 months after exacerbation will be evaluated by the actigraph (activPAL3TM - PAL Technologies Ltd., Glasgow, United Kingdom) through the number of steps, time spent in different positions during 7 days, 3 months after the first contact.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Di Lorenzo, PhD, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Special Respiratory Physiotherapy Unit of the Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler J, Malone D. Early mobilization in the intensive care unit: a systematic review. Cardiopulm Phys Ther J. 2012 Mar;23(1):5-13. PMID 22807649
- [Background] Alison JA, McKeough ZJ. Pulmonary rehabilitation for COPD: are programs with minimal exercise equipment effective? J Thorac Dis. 2014 Nov;6(11):1606-14. doi: 10.3978/j.issn.2072-1439.2014.07.45. PMID 25478201
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Bailey PH. The dyspnea-anxiety-dyspnea cycle--COPD patients' stories of breathlessness: "It's scary /when you can't breathe". Qual Health Res. 2004 Jul;14(6):760-78. doi: 10.1177/1049732304265973. PMID 15200799
- [Background] Banzett RB, Lansing RW, Brown R, Topulos GP, Yager D, Steele SM, Londono B, Loring SH, Reid MB, Adams L, et al. 'Air hunger' from increased PCO2 persists after complete neuromuscular block in humans. Respir Physiol. 1990 Jul;81(1):1-17. doi: 10.1016/0034-5687(90)90065-7. PMID 2120757
- [Background] Bergner M. Quality of life, health status, and clinical research. Med Care. 1989 Mar;27(3 Suppl):S148-56. doi: 10.1097/00005650-198903001-00012. PMID 2646487
- [Background] Borges RC, Carvalho CR. Physical activity in daily life in Brazilian COPD patients during and after exacerbation. COPD. 2012 Dec;9(6):596-602. doi: 10.3109/15412555.2012.705364. PMID 23244169
- [Background] Eaton T, Young P, Fergusson W, Moodie L, Zeng I, O'Kane F, Good N, Rhodes L, Poole P, Kolbe J. Does early pulmonary rehabilitation reduce acute health-care utilization in COPD patients admitted with an exacerbation? A randomized controlled study. Respirology. 2009 Mar;14(2):230-8. doi: 10.1111/j.1440-1843.2008.01418.x. PMID 19272084
- [Background] Fromer L, Cooper CB. A review of the GOLD guidelines for the diagnosis and treatment of patients with COPD. Int J Clin Pract. 2008 Aug;62(8):1219-36. doi: 10.1111/j.1742-1241.2008.01807.x. Epub 2008 Jun 28. PMID 18547365
- [Background] He M, Yu S, Wang L, Lv H, Qiu Z. Efficiency and safety of pulmonary rehabilitation in acute exacerbation of chronic obstructive pulmonary disease. Med Sci Monit. 2015 Mar 18;21:806-12. doi: 10.12659/MSM.892769. PMID 25783889
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Moy ML, Wayne PM, Litrownik D, Beach D, Klings ES, Davis RB, Yeh GY. Long-term Exercise After Pulmonary Rehabilitation (LEAP): Design and rationale of a randomized controlled trial of Tai Chi. Contemp Clin Trials. 2015 Nov;45(Pt B):458-467. doi: 10.1016/j.cct.2015.09.004. Epub 2015 Sep 8. PMID 26362690
- [Background] Nguyen HQ, Chu L, Amy Liu IL, Lee JS, Suh D, Korotzer B, Yuen G, Desai S, Coleman KJ, Xiang AH, Gould MK. Associations between physical activity and 30-day readmission risk in chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Jun;11(5):695-705. doi: 10.1513/AnnalsATS.201401-017OC. PMID 24713094
- [Background] Puhan MA, Spaar A, Frey M, Turk A, Brandli O, Ritscher D, Achermann E, Kaelin R, Karrer W. Early versus late pulmonary rehabilitation in chronic obstructive pulmonary disease patients with acute exacerbations: a randomized trial. Respiration. 2012;83(6):499-506. doi: 10.1159/000329884. Epub 2011 Aug 16. PMID 21846962
- [Background] Ramos EM, de Toledo-Arruda AC, Fosco LC, Bonfim R, Bertolini GN, Guarnier FA, Cecchini R, Pastre CM, Langer D, Gosselink R, Ramos D. The effects of elastic tubing-based resistance training compared with conventional resistance training in patients with moderate chronic obstructive pulmonary disease: a randomized clinical trial. Clin Rehabil. 2014 Nov;28(11):1096-106. doi: 10.1177/0269215514527842. Epub 2014 Mar 19. PMID 24647863
- [Background] Seymour JM, Moore L, Jolley CJ, Ward K, Creasey J, Steier JS, Yung B, Man WD, Hart N, Polkey MI, Moxham J. Outpatient pulmonary rehabilitation following acute exacerbations of COPD. Thorax. 2010 May;65(5):423-8. doi: 10.1136/thx.2009.124164. PMID 20435864
- [Background] Vaes AW, Garcia-Aymerich J, Marott JL, Benet M, Groenen MT, Schnohr P, Franssen FM, Vestbo J, Wouters EF, Lange P, Spruit MA. Changes in physical activity and all-cause mortality in COPD. Eur Respir J. 2014 Nov;44(5):1199-209. doi: 10.1183/09031936.00023214. Epub 2014 Jul 25. PMID 25063247